CLINICAL TRIAL: NCT04205292
Title: Cesarean Scar Pregnancy Managed by Dilatation and Evacuation (D&E) Versus Hysteroscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gabriele Saccone, Principal Investigator, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 298-19
Record Dates: First submitted 2019-12-15; First posted 2019-12-19 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Scar; Previous Cesarean Section
MeSH Terms: conditions — Cicatrix | interventions — Hysteroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dilatation and Evacuation (D&E) (Active Comparator): Women in this group will receive an in-patient treatment with Dilatation and Evacuation (D&E) after two doses of Methotrexate .
  Interventions: Procedure: hysteroscopic
- hysteroscopic surgery (Experimental): Women in this group will receive hysteroscopic surgery after two doses of Methotrexate .
  Interventions: Procedure: hysteroscopic

INTERVENTIONS:
Procedure: hysteroscopic — Women in the intervention group will receive an inpatient treatment with two-dose of Methotrexate followed by hysteroscopic resection under ultrasound guidance

SUMMARY:
Cesarean scar pregnancy (CSP) is a relative "new" type of ectopic pregnancy where the fertilized egg is implanted in the muscle or fibrous tissue of the scar after a previous cesarean section.

A recent review amounts almost 31 different treatment modalities for CSP. A broad spectrum of options represents a real challenge for the health care provider. The choice may be made among expectant management, medical treatment, local treatment and surgical approach, also combined together. There is insufficient evidence to recommend any one specific intervention over another for caesarean scar pregnancy. Future studies are needed to define the optimal management of pregnancy for caesarean section scars.

Thus, we aim to compare the success rate of two different treatment of CSP: the medical management by using two-dose of Methotrexate (MTX) followed by dilation and evacuation (D&E) compared to single dose of two-dose of Methotrexate followed by hysperoscopic approach.

DETAILED DESCRIPTION:
Cesarean scar pregnancy (CSP) is a relative "new" type of ectopic pregnancy where the fertilized egg is implanted in the muscle or fibrous tissue of the scar after a previous cesarean section. Since the first description of cesarean scar pregnancy in 1978, its frequency has increased dramatically due to the significant increase in the percentage of cesarean section and development of transvaginal (TV) ultrasonography (US). The overall incidence of CSP is 1 in 1,800 to 1 in 2,200 pregnancies, it means 0.05-0.04% of all pregnancies. In women after a cesarean section, the frequency of CSP is approximately 0.15%, which constitutes 6.1% of all ectopic pregnancies in patients after at least one cesarean operation. The risk factors that favour implantation in the CS scar are not well understood; therefore, there are no guidelines for the practicing physicians to determine the women at risk. Uterine surgery, anomalous healing of the scar, previous preterm CS without labour or a term elective CS, breech presentation at previous CS short intervals between the CSP and last pregnancy, last pregnancy ended with abortion may be some of the risk factors for CSP.

Although the 15% of CSPs remain undiagnosed, developed egographic techniques and several new US signs of CSP invasiveness are allowing ever better diagnoses. Cali et al. tested the hypothesis the relationship between the gestational sac of the CSP, previous caesarean scar and the anterior uterine wall can be used to predict the evolution of these cases. In order to do this, they propose a new sonographic sign, the "cross-over sign" (COS) . This echographic sign is reflected in the clinical presentation of the CSP, so we can divide the patients into two different groups: type I "endogenic type" characterized by the COS2 insertion, ance type II "exogenic type" characterized by COS1 insertion, the latter with worse outcomes in term of maternal morbidity and mortality.

A recent review amounts almost 31 different treatment modalities for CSP. A broad spectrum of options represents a real challenge for the health care provider. The choice may be made among expectant management, medical treatment, local treatment and surgical approach, also combined together. There is insufficient evidence to recommend any one specific intervention over another for caesarean scar pregnancy. Future studies are needed to define the optimal management of pregnancy for caesarean section scars.

Thus, we aim to compare the success rate of two different treatment of CSP: the medical management by using two-dose of Methotrexate (MTX) followed by dilation and evacuation (D&E) compared to single dose of two-dose of Methotrexate followed by hysperoscopic approach.

ELIGIBILITY:
Inclusion Criteria:

* Singleton gestations;
* 18 years to 50 years;
* Diagnosis of CSP;
* Gestational age ≤ 8 weeks and 6 days;
* Therapy with systemic Methotrexate 2-dose;
* Thickness of myometrial layer ≥2 mm.

Exclusion Criteria:

* Diagnosis of cervical pregnancy, aborting intrauterine pregnancy, or any other anomalous implantation site;
* Gestational age >8 weeks and 6 days;
* Heavy vaginal bleeding at the time of randomization;
* Women who did not received Methotrexate or received a single dose or a local dose;
* Thickness of myometrial layer <2 mm
* Women who are unconscious, ill, mentally handicapped;
* Women under the age of 18 years or over the age of 50 years.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 54 (Estimated)
Dates: Start 2019-12-23 (Actual); Primary Completion 2021-12-15 (Estimated); Study Completion 2022-01-15 (Estimated)

PRIMARY OUTCOMES:
success rate of treatment protocols, | resolution of scar pregnancy, day 7
  defined as no further treatment required until the complete resolution of the scar pregnancy.

SECONDARY OUTCOMES:
Further treatment required until the complete resolution of the scar pregnancy | resolution of scar pregnancy, day 7
  Further treatment required until the complete resolution of the CSP (repeat administration of methotrexate (MTX) and/or other surgical procedures),
histerectomy | resolution of scar pregnancy, day 7
  histerectomy
Maternal transfusion | resolution of scar pregnancy, day 7
  Maternal transfusion

CONTACTS AND LOCATIONS:
Locations (1):
- Gabriele Saccone, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No
no plan

REFERENCES:
- [Derived] Di Spiezio Sardo A, Zizolfi B, Saccone G, Ferrara C, Sglavo G, De Angelis MC, Mastantuoni E, Bifulco G. Hysteroscopic resection vs ultrasound-guided dilation and evacuation for treatment of cesarean scar ectopic pregnancy: a randomized clinical trial. Am J Obstet Gynecol. 2023 Oct;229(4):437.e1-437.e7. doi: 10.1016/j.ajog.2023.04.038. Epub 2023 May 3. PMID 37142075